CLINICAL TRIAL: NCT07333573
Title: A Single-arm, Open-label Phase I/II Study to Evaluate the Safety and Preliminary Efficacy of Hypoxia-Inducible CD73/AXL-Targeting CAR-T Cells (XW-LTH-03) in Patients With Advanced Gastric Cancer
Brief Title: A Hypoxia-Inducible CAR-T Cell Targeting AXL and CD73 for Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: SHANGHAI SINOBAY BIOTECHNOLOGY CO., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSGC-CD73AXL-CART
Record Dates: First submitted 2025-09-23; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XW-LTH-03 Infusion (Experimental)
  Interventions: Biological: XW-LTH-03 Infusion

INTERVENTIONS:
Biological: XW-LTH-03 Infusion — CD73/AXL-Targeting Hypoxia-Inducible CAR-T

SUMMARY:
This is a single-arm, open-label clinical study evaluating the safety and preliminary efficacy of a novel hypoxia-inducible, bispecific CD73/AXL-targeting CAR-T cell product, XW-LTH-03, in patients with stage IV gastric cancer (GC). The primary objective is to assess the safety and tolerability of XW-LTH-03 infusions. Secondary objectives include the evaluation of its antitumor efficacy and the characterization of its pharmacokinetic profile by measuring the in vivo expansion and persistence of the CAR-T cells. Exploratory analyses aim to identify potential biomarkers associated with clinical response and toxicity, as well as to investigate the cellular and molecular mechanisms underlying potential treatment resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, male or female.
2. Clinically judged as unresectable Stage IV gastric cancer that has progressed on or is intolerant to standard therapy, or patients who voluntarily forego standard therapy.
3. Patients must provide tumor tissue samples, with positive AXL and CD73 confirmed by immunohistochemical (IHC) staining at a central laboratory: AXL positivity rate ≥50% with staining intensity ≥++, and CD73 positivity rate ≥30% with staining intensity ≥+.
4. ECOG Performance Status score of ≤ 1.
5. Life expectancy of ≥ 3 months.
6. At least one measurable lesion (≥ 1 cm).
7. More than 4 weeks since the last failed treatment, and any toxicities from previous treatments must have recovered to Grade ≤ 1.
8. Adequate organ function and bone marrow reserve, as defined by the following laboratory values within a specified period before enrollment:

1. Hemoglobin (Hb) ≥ 90 g/L. 2. Absolute Neutrophil Count (ANC) ≥ 1.0 × 10^9/L. 3. Absolute Lymphocyte Count ≥ 0.5 × 10^9/L. 4. Platelet count ≥ 100 × 10^9/L. 5. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN).

6. Serum amylase and lipase ≤ 1.0 × ULN. 7. Total bilirubin ≤ 1.5 × ULN. 8. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (calculated by the Cockcroft-Gault formula).

9. Prothrombin Time (PT) or International Normalized Ratio (INR), and Partial Thromboplastin Time (PTT) < 1.5 × ULN. (Patients receiving warfarin or heparin anticoagulation therapy may be enrolled if no underlying abnormality in these parameters is suspected, but require close monitoring with at least weekly testing until INR is stable).

9. Adequate cardiac and pulmonary function. 10. Women of childbearing potential must have a negative pregnancy test within 7 days before treatment initiation. All subjects must agree to use effective contraception during the treatment period and for 1 year thereafter.

11. Voluntary signing of a written informed consent form, good compliance, and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Active, known, or highly suspected autoimmune disease.
2. Patients with brain metastases who have active central nervous system symptoms. (Note: Patients with brain metastases who completed radiotherapy at least 3 months prior to enrollment and remain asymptomatic from CNS disease may be eligible).
3. Active, uncontrolled systemic infection.
4. Receiving high-dose corticosteroids (>10 mg/day of methylprednisolone or equivalent doses of other corticosteroids) or other immunosuppressive therapy within 14 days prior to enrollment.
5. History of severe allergy to other monoclonal antibodies.
6. Intolerance or allergy to the investigational drug.
7. History of interstitial lung disease.
8. Evidence of organ failure:

   * Cardiac: Class III or IV heart failure (per NYHA or other applicable criteria).
   * Hepatic: Class C liver function as per Child-Pugh score.
   * Renal: Renal failure or uremia stage.
   * Pulmonary: Symptoms of severe respiratory failure.
   * Neurological: Impaired consciousness.
9. Active Hepatitis B (HBsAg positive with detectable HBV DNA), active Hepatitis C (HCV RNA positive), or HIV antibody positive.
10. History of organ transplantation.
11. Active gastrointestinal bleeding, or history of gastrointestinal bleeding within the past month.
12. History of drug abuse, or psychological/psychiatric disorders that may compromise compliance with the study.
13. Any unstable condition or situation that may jeopardize the patient's safety or compliance in the study.
14. Thyroid dysfunction.
15. Prior treatment with any form of adoptive T-cell therapy.
16. Currently receiving anticoagulant or antiplatelet therapy.
17. Major surgery or significant trauma within 4 weeks prior to enrollment.
18. History of other malignant tumors within the past 3 years.
19. Judged by the investigator as unsuitable for cell therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 3 months
Incidence of Dose-Limiting Toxicities (DLTs) | 3 months
Maximum Tolerated Dose (MTD) or Recommended Phase II Dose (RP2D) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China